CLINICAL TRIAL: NCT00006439
Title: Effects of Home Visits on Medication Adherence in Children and Youth With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Not Applicable | Model: Single Group | Purpose: Educational/Counseling/Training
Other Study IDs: NCRR-M01RR00069-0622; M01RR000069 (NIH)
Record Dates: First submitted 2000-11-04; First posted 2000-11-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Counseling

INTERVENTIONS:
Behavioral: Counseling in the home

SUMMARY:
Adherence to complex medication regimens is critical to successful treatment of HIV infection. Unfortunately, adherence to medical regimens with conventional interventions averages 50% in chronic disease. We have observed that adherence barriers that were unrecognized by providers in the clinic setting have been detected during home visits. It is possible that recognition and interventions to resolve adherence barriers observed during home visits may improve adherence. This proposal will test the hypothesis that home-visits which identify previously unrecognized adherence barriers and provide support and education will increase medication adherence among children and youth with HIV infection and improve the patient/health care provider relationship. Specific aims of the study are: 1. Determine the impact of a series of home-visits on adherence to medication regimens for HIV infected youth and children. 1a. Adherence to medical regimens will be assessed before and after the series of home-visits using a self-report questionnaire and Microelectronic Monitoring System (MEMS) or in-home pill count. 1b. For each of these measures a percentage of adherence will be calculated and compared from a baseline to after the final home visit and after the six month follow up period. 2. Assess the changes in patient satisfaction from baseline to after the home-visits using a questionnaire completed by the patient/family. 3. Incorporate a pilot study to assess the changes in the provider's knowledge of the patient's family characteristics and home circumstances relevant to adherence following the home visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* English speaking
* Live in Denver metro area
* Taking >=1 antiretroviral medication

Ages: 0 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McFarland, Principal Investigator
Locations (1):
- The Children's Hospital, Denver, Colorado, United States